CLINICAL TRIAL: NCT04114695
Title: Aortic Calcification and Central Blood Pressure in Patients With Chronic Kidney Disease
Acronym: ACCEPT
Status: Completed | Type: Observational
Sponsor: Central Jutland Regional Hospital (Other)
Responsible Party: Principal Investigator, Jakob Tobias Nyvad, M.D., PhD-student, Central Jutland Regional Hospital
Other Study IDs: VEK-nr 66842
Record Dates: First submitted 2019-08-14; First posted 2019-10-03 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Arterial Calcification; Kidney Diseases; Coronary Artery Disease; Aortic Calcification; Stroke; Vascular Diseases; Vascular Calcification
MeSH Terms: conditions — Kidney Diseases; Coronary Artery Disease; Stroke; Vascular Diseases; Vascular Calcification

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole Blood, Plasma, Urine
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Non-CKD (eGFR >60 ml/min/1.73 m2): Patients with renal function considered normal for age (eGFR >60 ml/min/1.73 m2) without proteinuria or structural kidney disease.
- CKD stage 3a (eGFR 45-59 ml/min/1,73 m2): Patients with CKD stage 3a (eGFR 45-59 ml/min/1,73 m2)
- CKD stage 3b (eGFR 30-44 ml/min/1,73 m2): Patients with CKD stage 3b (eGFR 30-44 ml/min/1,73 m2)
- CKD stage 4 (eGFR 15-29 ml/min/1,73 m2): Patients with CKD stage 4 (eGFR 15-29 ml/min/1,73 m2)
- CKD stage 5 (eGFR <15 ml/min/1,73 m2): Patients with CKD stage 5 (eGFR <15 ml/min/1,73 m2). 50% of these patients will be in dialysis, while the other 50% will be pre-dialysis patients.

SUMMARY:
Aim and background:

This study will seek to identify physiological and biochemical factors explaining and predicting a higher than expected central (aortic) blood pressure (BP) in patients with chronic kidney disease (CKD). The basic hypothesis of the study is that the degree of aortic calcification is an important component of elevated central BP, which, in turn, is important for the organ-damage and increased risk of cardiovascular disease associated with CKD.

Methods:

Adult patients with varying degrees of CKD undergoing scheduled coronary angiography (CAG) at Aarhus University Hospital will be included in this study.

During the CAG procedure, systolic and diastolic BP is determined in the ascending part of aorta by a calibrated pressure transducer connected to the fluid-filled CAG catheter.

Simultaneous with the registration of invasive aortic BP, estimation of central BP is performed using radial artery tonometry (SphygmoCor®), while a corresponding brachial BP is also measured.

Prior to the CAG, a non-contrast CT scan of aorta in its entirety will be performed to enable blinded quantification of calcification in the wall of aorta and coronary arteries.

Furthermore, echocardiography, resting BP measurement and a range of blood- and urine samples will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Patient referred for planned CAG at the Department of Cardiology, Aarhus University Hospital (AUH)
* eGFR constantly either >60 ml/min or <60 ml/min in at least 2 separate blood-sample measurements over at least 3 months.
* Signed informed consent-form.

Exclusion Criteria:

* Antihypertensive treatment changed within the last two weeks prior to the CAG.
* Severe aortic valve stenosis (<1 cm) as central hemodynamics may be altered
* Maximum number of patients in CKD-group already reached.
* Atrial fibrillation or other cardiac arrhythmia making radial Pulse Wave Analysis (PWA) estimations impossible.
* Known significant stenosis of a. subclavia or a. brachialis
* Bilateral arteriovenous-fistula (even if one or both of these have been surgically removed) as this may significantly affect the pulse-wave form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for CAG can be included in the study if they satisfy all inclusion criteria and do not meet any exclusion criteria.
  The study cohort will consist of:
  1. 160 patients with CKD at various stages based on estimated glomerular filtration rate (eGFR): 40 patients in stage 3a (eGFR 45-59 ml/min/1,73 m2), 40 patients in stage 3b (30-44 ml/min/1,73 m2), 40 patients in stage 4 (15-29 ml/min/1,73 m2) and 40 in stage 5 (<15 ml/min/1,73 m2). The stage 5 patients will be distributed between non-dialysis and dialysis patients.
  2. 40 patients with renal function considered normal for age (eGFR ≥60 ml/min/1.73 m2) without proteinuria or structural kidney disease.
Sampling Method: Non-Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
The difference between directly measured and estimated aortic (central) systolic blood pressure and the corresponding brachial systolic blood pressure | During the CAG-procedure
  Systolic arterial pressure will be determined in the ascending part of aorta using a calibrated pressure transducer connected to the CAG catheter. Simultaneous measurement with af Oscillometric BP-device (Microlife A2 Basic) will be conducted. The difference in mmHg will be calculated.
The degree of aortic calcification | CT-scan will be performed prior to CAG if logistically possible and no later than 3 weeks after CAG. All Agatston scoring will be completed when all patients have been included in the study during the summer of 2021.
  The degree of calcification in the wall of the ascending, arcus, descending and abdominal aorta will be measured with a non-contrast CT scan. Agatston-scoring will be applied on the CT images 2 cm after the aortic valve to the aortic bifurcation to ensure that aortic valve calcification is not included in the score. All Agatston scoring will be performed by a radiologist blinded to information on patient biochemical characteristics.
The difference between directly measured and estimated aortic (central) diastolic blood pressure and the corresponding brachial diastolic blood pressure. | During the CAG procedure
  Diastolic arterial pressure will be determined in the ascending part of aorta using a calibrated pressure transducer connected to the CAG catheter. Simultaneous measurement with af Oscillometric BP-device (Microlife A2 Basic) will be conducted. The difference in mmHg will be calculated.

SECONDARY OUTCOMES:
Association between Matrix Gla Protein (MGP) and aortic calcification | Analysis will be performed as batch-analysis at the end of inclusion of patients summer 2021
  To establish a deeper understanding of the pathogenesis of central arterial calcification in CKD, MGP, a novel biochemical marker of arterial calcification, will be collected and analysed in all patients.
Association between Calcification propensity score (T50test) and aortic calcification | Analysis will be performed as batch-analysis at the end of inclusion of patients summer 2021
  To establish a deeper understanding of the pathogenesis of central arterial calcification in CKD Calcification propensity score (T50test) will be collected and analysed in all patients.
Association between sRANKL (soluble receptor activator of nuclear factor kappa-B ligand) and aortic calcification | Analysis will be performed as batch-analysis at the end of inclusion of patients summer 2021
  To establish a deeper understanding of the pathogenesis of central arterial calcification in CKD sRANKL (soluble receptor activator of nuclear factor kappa-B ligand) will be collected and analysed in all patients.
Association between 25-OH-Vitamin D(D3+D2) and aortic calcification | Analysis will be performed as batch-analysis at the end of inclusion of patients summer 2021
  To establish a deeper understanding of the pathogenesis of central arterial calcification in CKD 25-OH-Vitamin D(D3+D2) will be collected and analysed in all patients.
Association between Fetuin-A(alfa-2-Heremans Schmid glycoprotein; AHSG) and aortic calcification | Analysis will be performed as batch-analysis at the end of inclusion of patients summer 2021.
  To establish a deeper understanding of the pathogenesis of central arterial calcification in CKD Fetuin-A(alfa-2-Heremans Schmid glycoprotein; AHSG) will be collected and analysed in all patients.
Association between Sclerostin and aortic calcification | Analysis will be performed as batch-analysis at the end of inclusion of patients summer 2021
  To establish a deeper understanding of the pathogenesis of central arterial calcification in CKD, Sclerostin will be collected and analysed in all patients.
Association between osteoprotegerin and aortic calcification | Analysis will be performed as batch-analysis at the end of inclusion of patients summer 2021
  To establish a deeper understanding of the pathogenesis of central arterial calcification in CKD, osteoprotegerin will be collected and analysed in all patients.
Association between BsAP (bone-specific alkaline phosphatase) and aortic calcification | Analysis will be performed as batch-analysis at the end of inclusion of patients summer 2021
  To establish a deeper understanding of the pathogenesis of central arterial calcification in CKD, BsAP (bone-specific alkaline phosphatase) will be collected and analysed in all patients.
Association between TRAP5B (tartrate-resistant acid phosphatase 5b) and aortic calcification | Analysis will be performed as batch-analysis at the end of inclusion of patients summer 2021
  To establish a deeper understanding of the pathogenesis of central arterial calcification in CKD, TRAP5B (tartrate-resistant acid phosphatase 5b) will be collected and analysed in all patients.
Association between P1NP (procollagen type 1 N propeptide) and aortic calcification | Analysis will be performed as batch-analysis at the end of inclusion of patients summer 2021
  To establish a deeper understanding of the pathogenesis of central arterial calcification in CKD, P1NP (procollagen type 1 N propeptide) will be collected and analysed in all patients.
Association between aortic calcification and Left Ventricular Global Longitudinal Strain (GLS) as determined during echocardiography. | No later than 1 month after central BP measurements
  All patients included in this study will undergo echocardiography. In particular systolic and diastolic function will be in focus. As scans will be supervised and reanalysed by a cardiologist blinded to patient CKD-stage.
Association between aortic calcification and LVDd (Left ventricular diameter in diastole) as determined during echocardiography. | No later than 1 month after central BP measurements
  All patients included in this study will undergo echocardiography. In particular systolic and diastolic function will be in focus. As scans will be supervised and reanalysed by a cardiologist blinded to patient CKD-stage.
Association between aortic calcification and IVS (Interventricular septum thickness) as determined during echocardiography. | No later than 1 month after central BP measurements
  All patients included in this study will undergo echocardiography. In particular systolic and diastolic function will be in focus. As scans will be supervised and reanalysed by a cardiologist blinded to patient CKD-stage.
Association between aortic calcification and Two-dimensional automated evaluation of ejection fraction (2-D auto-EF) as determined during echocardiography. | No later than 1 month after central BP measurements
  All patients included in this study will undergo echocardiography. In particular systolic and diastolic function will be in focus. As scans will be supervised and reanalysed by a cardiologist blinded to patient CKD-stage.
Association between aortic calcification and Aorta (sinus) diameter as determined during echocardiography. | No later than 1 month after central BP measurements
  All patients included in this study will undergo echocardiography. In particular systolic and diastolic function will be in focus. As scans will be supervised and reanalysed by a cardiologist blinded to patient CKD-stage.
Association between aortic calcification and Early mitral inflow velocity (E) as determined during echocardiography. | No later than 1 month after central BP measurements
  All patients included in this study will undergo echocardiography. In particular systolic and diastolic function will be in focus. As scans will be supervised and reanalysed by a cardiologist blinded to patient CKD-stage.
Association between aortic calcification and Duration of Pulmonal Vein Reversal as determined during echocardiography. | No later than 1 month after central BP measurements
  All patients included in this study will undergo echocardiography. In particular systolic and diastolic function will be in focus. As scans will be supervised and reanalysed by a cardiologist blinded to patient CKD-stage.
Association between aortic calcification and Late mitral inflow velocity (A) as determined during echocardiography. | No later than 1 month after central BP measurements
  All patients included in this study will undergo echocardiography. In particular systolic and diastolic function will be in focus. As scans will be supervised and reanalysed by a cardiologist blinded to patient CKD-stage.
Association between aortic calcification and Early diastolic mitral annulus velocity (E') as determined during echocardiography. | No later than 1 month after central BP measurements
  All patients included in this study will undergo echocardiography. In particular systolic and diastolic function will be in focus. As scans will be supervised and reanalysed by a cardiologist blinded to patient CKD-stage.
Association between aortic calcification and PW (Posterior wall thickness) as determined during echocardiography. | No later than 1 month after central BP measurements
  All patients included in this study will undergo echocardiography. In particular systolic and diastolic function will be in focus. As scans will be supervised and reanalysed by a cardiologist blinded to patient CKD-stage.
Association between aortic calcification and Aorta (ascendens) diameter as determined during echocardiography. | No later than 1 month after central BP measurements
  All patients included in this study will undergo echocardiography. In particular systolic and diastolic function will be in focus. As scans will be supervised and reanalysed by a cardiologist blinded to patient CKD-stage.
Association between aortic calcification and RVDd (Right ventricular diameter in diastole) as determined during echocardiography. | No later than 1 month after central BP measurements
  All patients included in this study will undergo echocardiography. In particular systolic and diastolic function will be in focus. As scans will be supervised and reanalysed by a cardiologist blinded to patient CKD-stage.
Association between aortic calcification and LAD (Left atrial diameter) as determined during echocardiography. | No later than 1 month after central BP measurements
  All patients included in this study will undergo echocardiography. In particular systolic and diastolic function will be in focus. As scans will be supervised and reanalysed by a cardiologist blinded to patient CKD-stage.
Association between aortic calcification and LAV (Left atrial volume) as determined during echocardiography. | No later than 1 month after central BP measurements
  All patients included in this study will undergo echocardiography. In particular systolic and diastolic function will be in focus. As scans will be supervised and reanalysed by a cardiologist blinded to patient CKD-stage.
Association between aortic calcification and TEI-Index as determined during echocardiography. | No later than 1 month after central BP measurements
  All patients included in this study will undergo echocardiography. In particular systolic and diastolic function will be in focus. As scans will be supervised and reanalysed by a cardiologist blinded to patient CKD-stage.
Association between aortic calcification and Tricuspid annular plane systolic excursion (TAPSE) as determined during echocardiography. | No later than 1 month after central BP measurements
  All patients included in this study will undergo echocardiography. In particular systolic and diastolic function will be in focus. As scans will be supervised and reanalysed by a cardiologist blinded to patient CKD-stage.
Association of arterial stiffness (defined as Pulse Wave Velocity (PWV)) and aortic calcification | No later than 1 month after Central BP.
  To get a non-invasive estimate of arterial stiffness, measurement of Pulse Wave Velocity (PWV) (carotid-femoral and carotid-radial) will be performed. PWV will be recorded with the Sphygmocor® device according to regular protocol. Calibration of the device will be performed using an oscillometric device after 5 minutes of rest. Only measurements with an estimated standard deviation of +/- 1.0 m/s will be accepted and included in the study. If possible, two acceptable measurements will be conducted for each included patient. Calculation of PWV will be performed automatically by the device using a previously published formula.

CONTACTS AND LOCATIONS:
Overall Officials: Niels H Buus, MD PhD DMSc, Study Chair — Department of Renal diseases, Aarhus University Hospital; Jakob T Nyvad, M.D., Principal Investigator — The Clinic of Hypertension, Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Derived] Nyvad J, Christensen KL, Andersen G, Reinhard M, Norgaard BL, Madsen JS, Nielsen S, Thomsen MB, Jensen JM, Peters CD, Buus NH. PIVKA-II but not dp-ucMGP is associated with aortic calcification in chronic kidney disease. BMC Nephrol. 2024 Nov 27;25(1):426. doi: 10.1186/s12882-024-03876-5. PMID 39604863
- [Derived] Nyvad J, Christensen KL, Andersen G, Reinhard M, Maeng M, Nielsen S, Thomsen MB, Jensen JM, Norgaard BL, Buus NH. Aortic Calcification is Associated With the Difference Between Invasive Central and Cuff-Measured Brachial Blood Pressure in Chronic Kidney Disease. Am J Hypertens. 2024 Jun 14;37(7):455-464. doi: 10.1093/ajh/hpae029. PMID 38477704